CLINICAL TRIAL: NCT05285787
Title: A Phase 2 Prospective Safety/Tolerability, Pharmacokinetics, Surrogate Biomarkers as Proxies for Efficacy Trial of EPN-701 in Subjects With Stable End Stage Renal Disease (ESRD) Receiving Outpatient Hemodialysis
Brief Title: A Clinical Trial of Epizon-701 (EPN-701) in Subjects With End-Stage Renal Disease (ESRD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Epizon Pharma, Inc. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EPN-701-001
Record Dates: First submitted 2022-02-16; First posted 2022-03-18 (Actual); Results first posted 2024-09-25 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-05

CONDITIONS: End-Stage Renal Disease (ESRD)
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — menaquinone 7

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- EPN-701, 10mg orally daily over 14 days (Experimental): Single arm
  Interventions: Drug: EPN-701 (Oral)

INTERVENTIONS:
Drug: EPN-701 (Oral) — MK-7
  Other Names: menaquinone-7

SUMMARY:
Patients with End Stage Renal Disease (ESRD) are prone to early and accelerated vascular calcification. Both the prevalence and extent of the vascular calcification are predictive for cardiovascular morbidity and all-cause mortality in this population. There is a growing body of evidence suggesting that dialysis patients have a primary, functional deficiency of Vitamin K2 as evidenced by reduced levels of circulating biomarkers including carboxylated forms of Matrix Gla Protein (MGP), Osteocalcin, and Fetuin-A, which are important inhibitors of vascular calcification. Decreased levels of Vitamin K2 are known to lead to microvascular calcification and are associated with dermatological and cardiovascular conditions such as calciphylaxis and peripheral arterial disease (PAD).

The purpose of this Phase 2 study is to examine the safety and pharmacokinetics of EPN-701 (menaquinone-7; MK-7) and to assess the effects on certain circulating biomarkers when MK-7 is orally administered once daily for 14 days.

DETAILED DESCRIPTION:
Patients with End Stage Renal Disease (ESRD) are prone to early and accelerated vascular calcification. Both the prevalence and extent of the vascular calcification are predictive for cardiovascular morbidity and all-cause mortality in this population. There is a growing body of evidence suggesting that dialysis patients have a primary, functional deficiency of Vitamin K2 as evidenced by reduced levels of circulating biomarkers including carboxylated forms of Matrix Gla Protein (MGP), Osteocalcin, and Fetuin-A, which are important inhibitors of vascular calcification. Decreased levels of Vitamin K2 are known to lead to microvascular calcification and are associated with dermatological and cardiovascular conditions such as calciphylaxis and peripheral arterial disease (PAD). The purpose of this Phase 2 study is to examine the safety and pharmacokinetics of EPN-701 (menaquinone-7; MK-7) and to assess the effects on certain circulating biomarkers when MK-7 is orally administered once daily for 14 days.

ELIGIBILITY:
Inclusion Criteria:

* Consenting subjects.
* Adult male and female who were diagnosed with stable ESRD.
* Subjects treated with maintenance hemodialysis at least 3 times a week for at least 3 months prior to the first dose of study drug.
* Clinically stable.

Exclusion Criteria:

* Solid organ transplant.
* Malignancy.
* Severe infection requiring intravenous (IV) antibiotics.
* Any co-existing disease or condition that could have compromised the safety of study participants and/or the integrity of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark T Smith, MD, Principal Investigator — Southeastern Clinical Research Institute, LLC 1521, Anthony Road Augusta, GA 30904
Locations (1):
- Southeastern Clinical Research Institute, LLC, Augusta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- EPN-701, 10mg Orally Daily Over 14 Days: Single arm
  EPN-701 (Oral): MK-7
  Over 14 days
Period: Overall Study
Arm/Group | EPN-701, 10mg Orally Daily Over 14 Days
Started | 18
Completed | 17
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | EPN-701, 10mg Orally Daily Over 14 Days
Number analyzed (Participants) | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 16
  >=65 years | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.4 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 18
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 18
Undercarboxylated Matrix Gla Protein (MGP), (pmol/L). [Mean (Standard Deviation); unit: pmol/L] | 1031.66 (422.563)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs)
Description: Number of Participants with:
  Treatment-emergent AEs Treatment-emergent AEs assessed as related to the study drug. Serious Adverse Events Deaths
Time Frame: Through study completion; over 14 days treatment and one week follow up.
Population: All patients who received at least one dose of EPN-701 was included in the safety evaluation.
Measure: Number; unit: participants
Groups:
- EPN-701 Treatment Arm: Participants who received study drug
Arm/Group | EPN-701 Treatment Arm
Number analyzed (Participants) | 18
participants | 8

2. Secondary Outcome: Plasma Concentrations of EPN-701.
Description: • Maximum plasma concentration of EPN-701 (Cmax) [ng/mL].
Time Frame: Through study completion; over 14 days treatment and one week follow-up.
Population: Pharmacokinetic (PK) Population: All enrolled patients who received all 14 days of dosing of study drug.
Measure: Mean (Standard Error); unit: ng/mL
Groups:
- Plasma Concentrations of EPN-701: Single arm
  EPN-701 (Oral): MK-7
Arm/Group | Plasma Concentrations of EPN-701
Number analyzed (Participants) | 15
ng/mL | 256 (138)

3. Secondary Outcome: Time to Maximum Plasma Concentration of EPN-701.
Description: Time to maximum plasma concentration of EPN-701 (Tmax) (h).
Time Frame: Through study completion; over 14 days treatment and one week follow-up.
Population: All enrolled patients who received all 14 days of dosing of study drug.
Measure: Mean (Standard Error); unit: hours
Arm/Group | Plasma Concentrations of EPN-701
Number analyzed (Participants) | 15
hours | 5.83 (1.66)

4. Other Pre Specified Outcome: Change From Baseline to Day 15 in Circulating Biomarker: Undercarboxylated Matrix Gla Protein (MGP), (Pmol/L).
Description: The percent change in circulating biomarker: Undercarboxylated MGP (pmol/L) levels from Day 1 (Baseline) to Day 15 was measured.
Time Frame: Day 1 to Day 15
Population: Patients who had evaluable biomarker levels at Day 1 and Day 15.
Measure: Mean (Standard Deviation); unit: percent change
Groups:
- Day 15 Biomarker Evaluation Group: Participants who had available Baseline and Day 15 measures of undercarboxylated MGP
Arm/Group | Day 15 Biomarker Evaluation Group
Number analyzed (Participants) | 18
percent change | -50.72 (20.041)

5. Other Pre Specified Outcome: Change From Baseline to Day 22 in Circulating Biomarker: Undercarboxylated Matrix Gla Protein (MGP), (Pmol/L).
Description: The percent change in circulating biomarker: Undercarboxylated MGP (pmol/L) levels from Day 1 (Baseline) to Day 22 was measured.
Time Frame: Day 1 to Day 22
Population: Patients who had evaluable biomarker levels at Day 1 and Day 22.
Measure: Mean (Standard Deviation); unit: percent change
Groups:
- Day 22 Biomarker Evaluation Group: Participants who had available Baseline and Day 22 measures of undercarboxylated MGP
Arm/Group | Day 22 Biomarker Evaluation Group
Number analyzed (Participants) | 17
percent change | -48.41 (19.994)

6. Other Pre Specified Outcome: Mean Value of Circulating Biomarker: Undercarboxylated Matrix Gla Protein (MGP), (Pmol/L) at Day 22.
Description: The mean value of circulating biomarker: Undercarboxylated MGP (pmol/L) levels on Day 22 was measured.
Time Frame: Day 22
Population: Patients who had evaluable biomarker levels at Day 1 and Day 22.
Measure: Mean (Standard Deviation); unit: pmol/L
Arm/Group | Day 22 Biomarker Evaluation Group
Number analyzed (Participants) | 17
pmol/L | 468.80 (143.733)

7. Other Pre Specified Outcome: Mean Measure of Circulating Biomarker: Undercarboxylated Matrix Gla Protein (MGP), (Pmol/L).
Description: Mean value of circulating biomarker: Undercarboxylated MGP (pmol/L) levels on Day 15 was measured.
Time Frame: Day 15
Population: Patients who had evaluable biomarker levels at Day 1 and Day 15.
Measure: Mean (Standard Deviation); unit: pmol/L
Arm/Group | Day 15 Biomarker Evaluation Group
Number analyzed (Participants) | 18
pmol/L | 439.32 (117.083)

ADVERSE EVENTS:
Time Frame: 14 days of treatment and 7 days of follow up.
Groups:
- Adverse Events (AEs): All patients who received at least one dose of study drug EPN-701 were included in the safety evaluation.
  (None of the Treatment Emergent Adverse Events were considered to be related to study drug.)
Arm/Group | Adverse Events (AEs)
All-Cause Mortality (participants affected / at risk) | 0/18
Serious Adverse Events (participants affected / at risk) | 2/18
Other Adverse Events (participants affected / at risk) | 8/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Adverse Events (AEs) (N=18)
cholelithiasis (Hepatobiliary disorders) | 1 — A patient experienced a serious adverse event of "cholelithiasis."
Pseudoaneurysm of Arteriovenous graft (Product Issues) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Adverse Events (AEs) (N=18)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1)
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Vascular graft complication (Injury, poisoning and procedural complications) | 1 (1) — Vascular Graft complication
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Peroneal nerve palsy (Nervous system disorders) | 1 (1) — Peroneal Nerve Palsy
Priapism (Reproductive system and breast disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) — Hypertension
Nausea (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Oedema peripheral (General disorders) | 1 (1)
Hyperkalaemia (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-01-16): https://cdn.clinicaltrials.gov/large-docs/87/NCT05285787/Prot_SAP_000.pdf